CLINICAL TRIAL: NCT03397004
Title: Doxycycline Crossover Trial for Hereditary Hemorrhagic Telangiectasia
Brief Title: Doxycycline for Hereditary Hemorrhagic Telangiectasia
Acronym: HHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Barrow Neurological Institute (Other); Duke University (Other); Feinstein Institute for Medical Research (Other); University of Pittsburgh (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 160517448; Award Number W81XWH-17-1-0429 (Other Grant/Funding Number: US Depart of Defense)
Record Dates: First submitted 2017-11-21; First posted 2018-01-11 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: Hereditary hemorrhagic telangiectasia; HHT; Doxycycline
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Doxycycline; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- doxycycline Hyclate (Active Comparator): subjects will be treated with a 6-month course of doxycycline oral capsule at a dose of 100mg twice daily
  Interventions: Drug: Doxycycline Hyclate
- Placebo (Placebo Comparator): subjects will be given a placebo oral capsule twice daily for 6-months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline Hyclate — Doxycycline will be given for 6 months, followed by a washout period for 6 months (pre or post a crossover intervention)
  Other Names: capsule
  Arms: doxycycline Hyclate
Drug: Placebo — Placebo will be given for 6 months, followed by a washout period for 6 months (pre or post a crossover intervention)
  Other Names: capsule
  Arms: Placebo

SUMMARY:
This study will investigate the effectiveness of oral doxycycline for the treatment of recurrent nasal hemorrhage in Hereditary Hemorrhagic Telangiectasia (HHT) subjects. The primary outcome for the trials will be the reduction of epistaxis severity (minutes of bleeding per week). The biological outcomes of interest are the regression of vascular malformations as well as tissue and circulation biomarkers of the relevant mechanistic pathways. A Phase II, randomized double-blind placebo-controlled crossover trial. Approximately 30 subjects with HHT, with moderate-severe recurrent epistaxis will participate in the randomized double-blind placebo-controlled cross over trial. Subject will be treated with a 6-month course of doxycycline 100mg twice daily or placebo twice daily.

DETAILED DESCRIPTION:
The aim is to study is to evaluate doxycycline as a treatment for HHT with the proposed "HHT Clinical Trial Protocol". Rare disease presents a number of challenges in clinical trial design, including recruitment challenges, related power limitations and less knowledge about outcomes measurement. Considering these limitations, as well as the large variability in epistaxis measures across HHT patients, a crossover-trial design, with each subject receiving the study drug and placebo, and therefore serving as their own control, has been selected, including randomization and blinding, to limit bias in measuring this subjective outcome.

This study will investigate doxycycline, given its demonstrated anti-angiogenic and anti-inflammatory properties, as well as compelling effects in arteriovenous malformation (AVM) models. Doxycycline also has the advantages of a proven safety track record for long-term use, oral administration and low cost. Doxycycline suppresses vascular endothelial growth factor (VEGF)-induced cerebral matric metalloproteinase-9 (MMP-9) activity in vivo in the mouse model, and has anti-inflammatory effects as well, via inhibition of pro-inflammatory cytokines. In human brain vascular malformation tissue, there is evidence of increased expression of MMP-9 and VEGF and another tetracycline, minocycline, has attenuated brain hemorrhage in the mouse. Recently, a small retrospective case series reported sustained reduction in nasal hemorrhage in seven HHT patients treated with oral doxycycline. We hypothesize that oral doxycycline will reduce nasal hemorrhage in HHT subjects, through anti-angiogenic and/or anti-inflammatory mechanisms, both of which have been implicated in HHT.

This is a double-blind randomized placebo-controlled trial (N=30) of oral doxycycline (100mg twice daily, 6-month course) in HHT subjects with moderate-severe recurrent nasal hemorrhage. Drug dosing and safety monitoring will be tailored specifically to the agent studied. The primary outcome will be reduction of bleeding minutes per week. In addition, vascular malformation tissue (cutaneous) will be obtained pre and post-treatment, and stained for inflammatory, angiogenic and bone morphogenetic protein-9 (BMP9)-activin A receptor like type1(ALK1)-endoglin- Smad1/5/9 pathway markers. In addition, pre-excision, vascular malformations will be imaged with speckle variance optical coherence tomography (SVOCT), in vivo non-invasive micro-angiography to measure lesion structure, vessel volume and vessel density, as previously described. If the drugs studied are effective at reducing nasal hemorrhage, this will have important clinical implications for HHT patients, and the tissue and imaging may provide important insights into mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age >+ 18 years
* Clinical HHT diagnosis or genetic diagnosis of HHT
* Known personal or familial endoglin (ENG), ALK1 or SMAD4 mutation
* Epistaxis at least 15 min per week (mean for past month)
* At least two skin telangiectases

  * >2mm diameter available for excisional biopsy,
  * at least two other telangiectases (skin or mucosal) available for micro-imaging
* Ability to give written informed consent

  * including compliance with the requirements of the study

Exclusion Criteria:

* Allergy/intolerance to the study drug or related agents
* Unstable medical illness
* Acute infection
* Creatinine > upper limit of normal (ULN)
* Liver transaminases (AST or ALT) >= 2x ULN
* Recent (within 2 month) use of study drug or other tetracycline agents
* Women who are pregnant
* Breastfeeding
* Plan to become pregnant during of the study
* Beta human chorionic gonadotropin (BHCG) level <6 IUL (re-test if 6-24 IU/L)
* Specific contra-indications for study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The reduction in epistaxis (nose bleeding) severity over 96 weeks | daily for 96 weeks
  Participants will be asked to maintain a daily diary for the duration of the study (96 weeks). Participants will record all epistaxis events daily, noting the duration in minutes and whether or not there was gushing during each nosebleed. The change in epistaxis severity will be measured from a sum of duration of all bleeding events each week, as measured from the participant daily diary.

SECONDARY OUTCOMES:
Change in epistaxis severity score (ESS) | baseline, week 12, week 24, week 36, week 48, week 60, week 72, week 84, week 96
  The epistaxis severity score is a six item questionnaire used to calculate a severity of HHT related nose bleeding. Each question is pertaining to the subject's typical symptoms within the last 3 months period. The first three questions are related to frequency, duration and intensity. The forth question whether or not medical attention was sought for nose bleeding. The remaining two questions are related to the presence of anemia and the need for blood transfusion due to nose bleeding. The resulting epistaxis severity score vary between; none 0-1, mild bleeding >1-4, moderate bleeding >4-7 and >7-10 for severe bleeding.
Measures related to chronic bleeding by a change from baseline | Baseline, week 12, week 18, week 24, week 30, week 36, week 42, week 48, week 60, week 66, week 72, week 78, week 84, week 96
  Blood samples will be taken to measure change in chronic bleeding by looking at the hemoglobin, ferritin and iron saturation level. Samples will be taken prior to investigational product for a baseline value. This will be followed by measurements every six weeks during the periods of investigational product for comparative analysis.
Regression of vascular malformations using Micro-imaging measures | week 12 (day 0), week 36, week 60, week 84
  Telangiectases will be micro-imaged using an established medical imaging technique speckle variance optical coherence tomography (SVOCT). The micro-imaging will be used for vasculature measurements. The SVOCT will measure the telangiectasia lesion area, volume, and density, lesion flow velocity and volume flow rate. Structural images will be generated. Imaging will be performed at four time points throughout the duration of the study.
Elucidate the mechanisms of action of doxycycline using tissue sample | week 36, week 84
  A punch biopsy of one cutaneous telangiectasia will be performed at two time points during the study. The biopsy tissue sample will be taken at the end of each 6 month active comparator (drug) or placebo treatment. The tissue will be analyze for lesion vessel density, distribution of vessel types (capillary, venule, arteriole) and for insights into mechanisms. Further investigation will include staining for inflammatory, angiogenesis and BMP9-ALK1-endoglin-Smad1/5/9 pathway markers (VEGF, MMP-9, cyclooxygenase-2 (COX-2), Endoglin, ALK1).
The measurement of a change in biomarkers | week 12 (day 0), week 24, week 36, week 48, week 60, week 72, week 84, week 96
  Serum, plasma levels will be measured for inflammatory, angiogenic, and BMP9-ALK1-endoglin-Smad1/5/9 pathway (VEGF, MMP-9, Thrombospondin-2, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), endothelin). Biomarker samples will be collected every 3-months. This will allow each subject to also provide their own controls for each treated case. The change in biomarkers will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Faughnan, MD MSc FRCPC, Principal Investigator — St. Michael's Hospital / The University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson KP, Sykes J, Chandakkar P, Marambaud P, Vozoris NT, Marchuk DA, Faughnan ME. Randomized, double-blind, placebo-controlled, crossover trial of oral doxycycline for epistaxis in hereditary hemorrhagic telangiectasia. Orphanet J Rare Dis. 2022 Nov 7;17(1):405. doi: 10.1186/s13023-022-02539-8. PMID 36344987